CLINICAL TRIAL: NCT01458873
Title: Intravenous Sodium Bicarbonate Verifies Intravenous Position of Catheters in Spontaneously Breathing Adult Volunteers
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Ilan Keidan, Director, Pediatric Anesthesia, Sheba Medical center, Sheba Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: SHEBA-11-8716-IK-CTIL
Record Dates: First submitted 2011-10-09; First posted 2011-10-25 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: Infiltration; Extravasation
Keywords: infiltration; extravasation
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- sodium bicarbonate 4.2% (Experimental): sodium bicarbonate 4.2% 50 m"l
  Interventions: Drug: sodium bicarbonate 4.2%
- sodium bicarbonate 2.1% (Experimental): sodium bicarbonate 2.1% 1 50 m"l
  Interventions: Drug: diluted sodium bicarbonate 2.1%
- normal saline (Placebo Comparator): 50 m"l normal saline
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: sodium bicarbonate 4.2% — diluted sodium bicarbonate 50 ml
  Arms: sodium bicarbonate 4.2%
Drug: diluted sodium bicarbonate 2.1% — 50ml
  Other Names: sodium bicarbonate 2.1%
  Arms: sodium bicarbonate 2.1%
Drug: normal saline — 50ml
  Arms: normal saline

SUMMARY:
Vascular access in patients carries a significant risk of accidental extravasation of intravenous (IV) fluids and medications with the potential for tissue injury. This prospective controlled study assessed the diagnostic utility of using intravenous diluted sodium bicarbonate to confirm placement of IV catheters in volunteers . Diluted sodium bicarbonate or 0.9% normal saline, will be injected in a randomized order while end-tidal carbon dioxide in the exhaled air will be monitored. The investigators hypothesize that the injected bicarbonate will dissolve into carbon dioxide and water and cause a transient increase in the measured exhaled CO2.

The effect is unique to bicarbonate and will not appear once normal saline is injected. the safety of the administration of bicarbonate on the metabolic profile of the volunteers will be assessed by measurement of venous blood pH and electrolytes.

DETAILED DESCRIPTION:
Vascular access in patients carries a significant risk of accidental extravasation of intravenous (IV) fluids and medications with the potential for tissue injury. This prospective controlled study assessed the diagnostic utility of using intravenous diluted sodium bicarbonate to confirm placement of IV catheters in volunteers . Diluted sodium bicarbonate or 0.9% normal saline, will be injected in a randomized order while end-tidal carbon dioxide in the exhaled air will be monitored. The investigators hypothesize that the injected bicarbonate will dissolve into carbon dioxide and water and cause a transient increase in the measured exhaled CO2. Arbitrary increase of more than 10%in end-tidal carbon dioxide is considered as a positive response.

The effect is unique to bicarbonate and will not appear once normal saline is injected. the safety of the administration of bicarbonate on the metabolic profile of the volunteers will be assessed by measurement of venous blood pH and electrolytes.

ELIGIBILITY:
Inclusion Criteria:

* ASA I,II
* no cardiovascular or respiratory disease

Exclusion Criteria:

* ASA > II
* Cardiovascular disease
* Respiratory disease
* renal failure
* metabolic alkalosis

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
transient increase in end tidal carbon dioxide | 4-12 seconds
  Once sodium bicarbonate is injected the measured end-tidal carbon dioxide will transiently increase by at least 10% of baseline

SECONDARY OUTCOMES:
Change in venous blood pH | 10-20 minutes
  Blood pH and will be measured prior and ten minutes after the injections
Subjective adverse symptoms associated with injection of sodium bicarbonate | 1 minute
  The subjective symptoms as well as hemodynamic changes associated with the injection of sodium bicarbonate will be recorded
change in venous blood sodium | 10- 20 minutes
  blood sodium level will be measured before and 10-20 minutes after the end of the injections.
change in venous blood bicarbonate level | 10-20 minutes
  blood level of bicarbonate will be measured before and 10-20 minutes after the injection.
change in venous blood potasium level | 10-20 minutes
  venous blood potasium level will be measured before and 10-20 minutes after injection

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Background] Keidan I, Ben-Menachem E, Barzilai A, Nur I, Berkenstadt H. Intravenous sodium bicarbonate verifies intravenous position of catheters in ventilated patients. Anesth Analg. 2011 Aug;113(2):279-81. doi: 10.1213/ANE.0b013e3182222ed0. Epub 2011 Jun 3. PMID 21642603
- [Derived] Keidan I, Sidi A, Ben-Menachem E, Derazne E, Berkenstadt H. A simple diagnostic test to confirm correct intravascular placement of peripheral catheters in order to avoid extravasation. J Clin Anesth. 2015 Nov;27(7):585-8. doi: 10.1016/j.jclinane.2015.07.004. Epub 2015 Aug 15. PMID 26286133